CLINICAL TRIAL: NCT00947037
Title: An Open-Label, Multi-Center, Follow-Up Study Designed to Evaluate the Long-Term Effects of AP-CD/LD in Fluctuating Parkinson's Disease Subjects
Brief Title: Gastric Retentive Carbidopa/ Levodopa in Parkinson's Patients; a One Year, Open Label, Safety Extension Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to postpone the performance of this study to after phase 3
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN 12 005
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extension (Experimental): Open label extension, 1 arm
  Interventions: Drug: AP-CD/LD

INTERVENTIONS:
Drug: AP-CD/LD

SUMMARY:
An extension of study IN 09 004 testing the long term safety of the Accordion Pill Carbidopa/Levodopa (AP-CD/LD)

ELIGIBILITY:
Inclusion Criteria:

* Subject satisfactorily completed study IN 09 004 and, in the opinion of the investigator, will benefit from participation in the extension study
* Subject with Parkinson's disease experiencing predictable motor fluctuations, end of dose "wearing off", defined by the patient's report of at least two episodes daily of a decline in function from peak benefit, with at least 2 hours OFF a day at the discretion of the PI (does not include early morning akinesia or nocturnal akinesia)
* Subject that has been treated for at least 3 months prior to the study with 500-1000 mg Levodopa + DDCI, in 4 or more divided doses per day
* Hoehn and Yahr stages I-III
* Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study
* Prepared and able to give written (signed and dated) informed consent, which includes compliance with study requirements and restrictions prior to admission to the study.

Exclusion Criteria

* Subject has undergone Deep brain stimulation (DBS) or any other neurological surgical procedure that affects neurological symptoms (e.g tremor, rigidity, stiffness, slowed movement, and walking problem)
* Subjects with any gastrointestinal surgery other than appendectomy or herniotomy, recent history of inflammatory bowel disease, irritable bowel syndrome, severe gastrointestinal narrowing, intestinal obstruction, or frequent nausea or emesis or diarrhea which, in the opinion of the investigator, contraindicates his/her participation
* Subjects with a recent history of clinically defined GERD, peptic ulcer or any gastrointestinal disorder likely to influence drug absorption which, in the opinion of the investigator, contraindicates his/her participation

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To assess patient and investigator global evaluation of, and degree of satisfaction with, AP-CD/LD (CGI, GSS)

SECONDARY OUTCOMES:
Quality of Life questionnaires
Daytime sleepiness
Efficacy measures of motor symptoms

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - TASMC, Tel Aviv